CLINICAL TRIAL: NCT03425591
Title: A Retro-Prospective Observational Study of Ibrutinib Treatment of Chronic Lymphocytic Leukemia and Mantle-cell Lymphoma in Routine Clinical Practice
Brief Title: A Study of Ibrutinib in the Treatment of Chronic Lymphocytic Leukemia and Mantle-cell Lymphoma in Routine Clinical Practice
Acronym: FIRE
Status: Completed | Type: Observational
Sponsor: Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR107363; 54179060CAN4001 (Other: Janssen-Cilag Ltd.)
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2022-10-06 (Actual); Status verified 2022-10

CONDITIONS: Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Mantle-Cell | interventions — ibrutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort 1: Chronic Lymphocytic Leukemia (CLL) Participants: Participants with confirmed diagnosis of CLL will be observed to collect data on ibrutinib therapy to describe the effectiveness of ibrutinib and to provide a description of ibrutinib therapy and the first non-ibrutinib subsequent therapy in Cohort 1. The primary data source for this observational study will be the medical records of each enrolled participant.
  Interventions: Drug: Ibrutinib
- Cohort 2: Mantle-Cell Lymphoma (MCL) Participants: Participants with confirmed diagnosis of MCL will be observed to collect data on ibrutinib therapy to describe the effectiveness of ibrutinib and to provide a description of ibrutinib therapy and the first non-ibrutinib subsequent therapy in Cohort 2. The primary data source for this observational study will be the medical records of each enrolled participant.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Participants in this observational study with confirmed diagnosis of CLL and MCL receiving ibrutinib in routine clinical practice settings will be observed for 5 years.

SUMMARY:
The purpose of this study is to describe the effectiveness of ibrutinib and to provide a description of ibrutinib therapy and the first non-ibrutinib subsequent therapy for chronic lymphocytic leukemia (CLL) and mantle-cell lymphoma (MCL).

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed diagnosis of chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL) or mantle-cell lymphoma (MCL), and is initiating ibrutinib therapy or has initiated ibrutinib therapy on or after 21 November 2014 (date of ibrutinib commercialization) for:

  1. treatment of CLL/SLL in participants who have received at least 1 prior therapy; or
  2. treatment in first line CLL/SLL participants in the presence of deletion (del) 17p or TP53 mutation in participants unsuitable for chemo-immunotherapy; or
  3. treatment of participants with relapsed or refractory MCL
* Not currently participating in another investigational study, clinical study, or any expanded access program at study entry
* Has not participated in the ibrutinib Autorisation Temporaire d'Utilisation (ATU) program
* Participant must sign a written informed consent form (ICF) allowing data collection and source data verification

Exclusion Criteria:

* Currently participating in another investigational study, clinical study, or any expanded access program at study entry
* Participated in the ibrutinib Autorisation Temporaire d'Utilisation (ATU) program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population include chronic lymphocytic leukemia (CLL) or mantle-cell lymphoma (MCL) participants who were or will be treated by ibrutinib per routine clinical care on or after 21 November 2014.
Sampling Method: Non-Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Progressive-Free Survival (PFS) | Approximately up to 5 years
  PFS in Chronic Lymphocytic Leukemia (CLL) and Mantle-Cell Lymphoma (MCL) participants will be determined. PFS is defined as the time from start of ibrutinib therapy to Progressive Disease (PD) or death from any cause. PD is defined as any new lesions or increase by greater than or equal to (>=) 50 percent (%) of previously involved sites from nadir.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Approximately up to 5 years
  ORR observed in CLL and MCL participants will be reported. ORR is defined as the proportion of participants with at least an objective response (that is, complete response or partial response, or partial response with lymphocytosis for CLL participants) as assessed by the participating physician.
Time to First Response | Approximately up to 5 years
  Time to First Response in CLL and MCL participants will be reported. Time to first response is defined as the time from start of ibrutinib therapy until first objective response.
Time to Best Response | Approximately up to 5 years
  Time to best response in CLL and MCL participants will be reported. Time to best response is defined as the time from start of ibrutinib therapy until best objective response.
Duration of Response | Approximately up to 5 years
  Duration of response in CLL and MCL participants will be reported. Duration of response is defined as the time from start of ibrutinib therapy until PD or death resulting from progression. PD is defined as any new lesions or increase by >=50% of previously involved sites from nadir.
Overall survival (OS) | Approximately up to 5 years
  Overall survival in CLL and MCL participants will be reported. Overall survival will be measured from start of ibrutinib therapy to the date of death (all-cause mortality); and from diagnosis to the date of death.
Duration of Ibrutinib Therapy | Approximately up to 5 years
  Duration of ibrutinib therapy in CLL and MCL participants will be reported.
Duration of a Treatment-Free Period | Every 6 months (Approximately up to 5 years)
  Duration of treatment-free period in CLL and MCL participants will be reported.
Duration of the First Non-Ibrutinib Subsequent Therapy Period | Approximately up to 5 years
  Duration of the first non-ibrutinib subsequent therapy period in CLL and MCL participants will be reported.
Participants' Daily Dose | Approximately up to 5 years
  Daily dose of ibrutinib taken by CLL and MCL participants will be analyzed.
Number of Participants Who Require Dose Modifications | Approximately up to 5 years
  Number of CLL and MCL participants requiring dose modifications in the ibrutinib therapy will be reported.
Number of Medications Added | Approximately up to 5 years
  Number of medications added in the CLL and MCL treatment will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Ltd. Clinical Trial, Study Director — Janssen-Cilag Ltd.
Locations (1):
- Paris, France

REFERENCES:
- [Derived] Dartigeas C, Quinquenel A, Ysebaert L, Dilhuydy MS, Anglaret B, Slama B, Le Du K, Tardy S, Tchernonog E, Orfeuvre H, Voillat L, Guidez S, Malfuson JV, Dupuis S, Deslandes M, Feugier P, Leblond V; FIRE Investigators Group. Final results on effectiveness and safety of Ibrutinib in patients with chronic lymphocytic leukemia from the non-interventional FIRE study. Ann Hematol. 2025 Feb;104(2):1079-1093. doi: 10.1007/s00277-024-05666-3. Epub 2024 Mar 6. PMID 38443660
- [Derived] Dartigeas C, Slama B, Doyle M, Tapprich C, Albrecht C, Dupuis S, Wapenaar R, Schmidt-Hieber C, Leblond V. FIRE Study: Real-World Effectiveness and Safety of Ibrutinib in Clinical Practice in Patients with CLL and MCL. Clin Hematol Int. 2022 Sep;4(3):65-74. doi: 10.1007/s44228-022-00015-5. Epub 2022 Sep 14. PMID 36103041